CLINICAL TRIAL: NCT01049009
Title: The Effect of Nebivolol on Endothelial Dysfunction in African Americans With Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00017946
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: High Blood Pressure
Keywords: Nitric Oxide; Adrenergic beta-Antagonists; Antihypertensive Agents; Vasodilator Agents; Anti-Arrhythmia Agents; Sympatholytics; Vascular Resistance; Neurotransmitter Agents; Cardiovascular Diseases; Metoprolol succinate; Therapeutic Uses; Metoprolol; Vascular Diseases; Nebivolol; Cardiovascular Agents; Endothelium-Dependent Relaxing Factors
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Vascular Diseases | interventions — Nebivolol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebivolol followed by Metoprolol XL (Active Comparator): Subjects are randomized to Nebivolol 5mg and titrate to Nebivolol 10mg two weeks after drug initiation. Ten weeks after titration subjects will cross over to Metoprolol XL 50mg and titrate to Metoprolol XL 100mg two weeks after cross over.
  Interventions: Drug: Nebivolol; Drug: Metoprolol XL
- Metoprolol XL followed by Nebivolol (Active Comparator): Subjects are randomized to Metoprolol XL 50mg and titrate to Metoprolol XL 100mg two weeks after drug initiation. Ten weeks after titration subjects will cross over to Nebivolol 5mg and titrate to Nebivolol 10mg two weeks after cross over.
  Interventions: Drug: Nebivolol; Drug: Metoprolol XL

INTERVENTIONS:
Drug: Nebivolol — Subjects will be randomized to either nebivolol or metoprolol xl, and remain on the study drug for 10 weeks. They will then "cross over" to take 10 weeks of the comparator drug.
Drug: Metoprolol XL — Subjects will be randomized to either nebivolol or metoprolol xl, and remain on the study drug for 10 weeks. They will then "cross over" to take 10 weeks of the comparator drug.

SUMMARY:
High blood pressure (hypertension) is called the "silent killer" because many people do not know they have it, and do not know when it is well controlled. Unfortunately, over time uncontrolled hypertension can cause irreversible organ damage that can lead to heart attack, stroke, heart failure, and kidney failure. If a person cannot control their blood pressure with diet and exercise, doctors often prescribe medications to help control the blood pressure. Nebivolol is a medication that has been recently approved by the FDA for the treatment of hypertension. Our study will investigate whether treatment with nebivolol, as compared to another medication called metoprolol, in African Americans with hypertension will be more effective in protecting blood vessels against the harmful effects of high blood pressure.

Over time high blood pressure causes hardening of the arteries (atherosclerosis) which leads to narrowing of the blood vessels and reduces blood flow to our organs. Arteries also relax and contract naturally, which further changes the blood supply. When arteries are narrowed, exercise can bring on a condition in which the blood supply is inadequate, and this might result in the sensation of pain.

Cells lining our blood vessels produce a variety of substances that normally cause arteries to relax. Two of these substances are called nitric oxide (NO) and endothelium-derived hyperpolarizing factor (EDHF). We are trying to determine the nature of these substances in African Americans with high blood pressure and how it is affected by nebivolol and metoprolol. One way to determine this is to inject drugs such as L-NMMA (N(G)-monomethyl-L-arginine) or TEA (tetraethylammonium chloride), which block the production of NO and EDHF respectively, and then study what happens to the blood flow at rest and during exercise. It is our thought that nebivolol, in comparison to metoprolol, will increase the substances that naturally cause arteries to relax and improve blood supply.

ELIGIBILITY:
Inclusion Criteria:

* Male or post-menopausal females aged 18-80 years.
* Subjects self-identified as black or African-American.
* Diagnosis of hypertension.
* Patients on current anti-hypertensive therapy that does not include beta blockade should have BP >135/85.
* Patients on anti-hypertensive therapy including beta blockers will have their beta blockers discontinued gradually over 2 weeks before enrolment.
* Concomitant therapy: Patients will be allowed to be on concomitant therapy with aspirin, statins, thiazide diuretics, calcium antagonists (for treatment of hypertension), clonidine, or vasodilators. Patients will be on stable medical therapy for at least 2 months before recruitment. Patients with previous treatment with beta adrenergic blockers (metoprolol, propranolol, atenolol, and labetalol) will also be eligible to participate, but will be randomized to the study beta blocker.

Exclusion Criteria:

* Initiation or change in dose of statin or other anti-hypertensive therapy within 2 months before the study
* Inability to return to Emory for follow-up testing
* Age < 21 or >80 years
* Premenopausal females with potential for pregnancy
* Acute infection in previous 2 weeks
* On angiotensin antagonists (ACE inhibitors or ARBs)
* History of substance abuse
* Current neoplasm
* Chronic renal failure [creatinine > 2.5 mg/dL] or liver failure (liver enzymes >2X normal)
* Acute coronary syndrome, Class IV heart failure, CVA, coronary intervention within 2 months
* Known aortic stenosis, hypertrophic cardiomyopathy.
* Inability to give informed consent

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Result] Neuman RB, Hayek SS, Poole JC, Rahman A, Menon V, Kavtaradze N, Polhemus D, Veledar E, Lefer DJ, Quyyumi AA. Nitric Oxide Contributes to Vasomotor Tone in Hypertensive African Americans Treated With Nebivolol and Metoprolol. J Clin Hypertens (Greenwich). 2016 Mar;18(3):223-31. doi: 10.1111/jch.12649. Epub 2015 Aug 19. PMID 26285691
- Available data/document: Publication: 26285691 — https://www.ncbi.nlm.nih.gov/pubmed/26285691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from the general medical clinics of The Emory Clinic, Emory University Hospital, and Grady Memorial Hospital between January 2010 through January 2012.
Pre-assignment Details: 91 subjects were enrolled but 47 subjects were withdrawn prior to group assignment due to various factors, which included eligibility criteria, lost to follow-up, and withdrawal by subject.
Groups:
- Nebivolol/Metoprolol XL: Subjects are randomized to Nebivolol 5mg and titrate to Nebivolol 10mg two weeks after drug initiation. Ten weeks after titration subjects will cross over to Metoprolol XL 50mg and titrate to Metoprolol XL 100mg two weeks after cross over.
- Metoprolol XL/Nebivolol: Subjects are randomized to Metoprolol XL 50mg and titrate to Metoprolol XL 100mg two weeks after drug initiation. Ten weeks after titration subjects will cross over to Nebivolol 5mg and titrate to Nebivolol 10mg two weeks after cross over.
Period: Treatment Period 1 (12 Weeks)
Arm/Group | Nebivolol/Metoprolol XL | Metoprolol XL/Nebivolol
Started | 23 | 21
Completed | 21 | 18
Not Completed | 2 | 3
Not completed — Protocol Violation | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Period: Treatment Period 2 (12 Weeks)
Arm/Group | Nebivolol/Metoprolol XL | Metoprolol XL/Nebivolol
Started | 21 | 18
Completed | 11 | 8
Not Completed | 10 | 10
Not completed — Lost to Follow-up | 2 | 3
Not completed — Protocol Violation | 8 | 7

BASELINE CHARACTERISTICS:
Population: Baseline population characteristics only account for subjects that completed the entire study.
Groups:
- Nebivolol/Metoprolol XL: Subjects were randomized to Nebivolol 5mg and titrated to Nebivolol 10mg two weeks after drug initiation. Ten weeks after titration, subjects crossed over to Metoprolol XL 50mg and titrated to Metoprolol XL 100mg two weeks after cross over.
- Metoprolol XL/Nebivolol: Subjects were randomized to Metoprolol XL 50mg and titrated to Metoprolol XL 100mg two weeks after drug initiation. Ten weeks after titration, subjects crossed over to Nebivolol 5mg and titrated to Nebivolol 10mg two weeks after cross over.
- Total: Total of all reporting groups
Arm/Group | Nebivolol/Metoprolol XL | Metoprolol XL/Nebivolol | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Function Measured by Forearm Blood Flow (FBF) at 12 Weeks
Description: Forearm blood flow measured by venous occlusion plethysmography at rest, after administration of N(G)-monomethyl-L-arginine (L-NMMA) and tetraethylammonium chloride (TEA), after administration of L-NMMA, TEA, and acetylcholine, and after administration of L-NMMA, TEA, and exercise. Unit of Measure refers to volume of blood (mL) per 100 mL of forearm tissue per minute.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mL/100 mL/min
Arm/Group | Nebivolol/Metoprolol XL | Metoprolol XL/Nebivolol
Number analyzed (Participants) | 11 | 8
mL/100 mL/min
  At rest | 2.739 (1.365) | 2.679 (.0901)
  L-NMMA+TEA | 1.963 (0.968) | 2.221 (0.630)
  L-NMMA+TEA+ACh | 5.376 (3.362) | 7.562 (4.358)
  L-NMMA+TEA+exercise | 7.377 (2.754) | 11.574 (4.716)

2. Primary Outcome: Endothelial Function Measured by Forearm Blood Flow (FBF) at 24 Weeks
Description: as for outcome 1
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: mL/100 mL/min
Arm/Group | Nebivolol/Metoprolol XL | Metoprolol XL/Nebivolol
Number analyzed (Participants) | 11 | 8
mL/100 mL/min
  At rest | 3.066 (1.469) | 2.968 (1.164)
  L-NMMA+TEA | 2.457 (1.549) | 2.287 (0.693)
  L-NMMA+TEA+ACh | 7.158 (4.875) | 7.534 (4.523)
  L-NMMA+TEA+exercise | 9.589 (3.550) | 10.395 (2.687)

ADVERSE EVENTS:
Description: Only subjects that were randomized into an arm with drug were included in the "at-risk participant" fields.
Arm/Group | Nebivolol/Metoprolol XL | Metoprolol XL/Nebivolol
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/21
Other Adverse Events (participants affected / at risk) | 0/23 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No